CLINICAL TRIAL: NCT01322698
Title: Staging Candidiasis in ICU Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2009/BL-01; 2010-A00858-31 (Other: ANSM)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Candidiasis
Keywords: ICU
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The target population includes patients in ICUs at the Nîmes and Montpellier University hospitals. This is a population of non-neutropenic patients (polynuclear neutrophils > 500/mm3) at risk of developing invasive candidiasis.
  Interventions: Biological: Tests for candidiasis

INTERVENTIONS:
Biological: Tests for candidiasis — Tests include (1) anti-candida antibody ELISA kit; (2) candida antigen ELISA kit; (3) detection of circulating Candida DNA via SYBR Breen qPCR Master mix; (4) colonization index based on mycological examination of five out of the following: urine, oral swab, bronchial aspirate, anal swab, swab of a central venous line, gastric liquid.

SUMMARY:
Our primary objective is to evaluate the relevance of the early determination of Candida infection status among non-neutropenic patients hospitalized over 48 hours in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Polynuclear neutrophils > 500/mm^3
* Hospitalized for > 48 hours in participating ICUs

Exclusion Criteria:

* Patients discharged from ICU in < 48h
* Patient diagnosed with invasive candidosis before entry to ICU
* Patient is taking an anti-fungal treatment
* polynuclear neutrophils < 500/mm^3
* patient transferred to another ICU
* patient included in the Abmidex protocole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes patients in ICUs at the Nîmes and Montpellier University hospitals. This is a population of non-neutropenic patients (polynuclear neutrophils > 500/mm3) at risk of developing invasive candidiasis.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10-07 (Actual); Study Completion 2014-10-07 (Actual)

PRIMARY OUTCOMES:
Number of positive Candidiasis tests | 7 days
  Number of tests (score of 0 to 4) positive for Candida. Tests include (1) anti-candida antibody ELISA kit; (2) candida antigen ELISA kit; (3) detection of ciruclating Candida DNA via SYBR Breen qPCR Master mix; (4) colonization index based on mycological examination of five out of the following: urine, oral swab, bronchial aspirate, anal swab, swab of a central venous line, gastric liquid.

SECONDARY OUTCOMES:
Number of positive Candidiasis tests | 2 days
  Number of tests (score of 0 to 4) positive for Candida. Tests include (1) anti-candida antibody ELISA kit; (2) candida antigen ELISA kit; (3) detection of ciruclating Candida DNA via SYBR Breen qPCR Master mix; (4) colonization index based on mycological examination of five out of the following: urine, oral swab, bronchial aspirate, anal swab, swab of a central venous line, gastric liquid.
Patient leaves ICU unit, yes/no | 1 month
Patient passes away in ICU unit, yes/no | 1 month
Patient has been prescribed an antifungal treatment in the past month, yes/no | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Lachaud, MD, Study Director — Centre Hospitalier Universitaire de Nîmes; Nathalie Bourgeois, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Nîmes, Nîmes, Gard
  - CHU de Montpellier, Montpellier

REFERENCES:
- [Result] Larcher R, Platon L, Amalric M, Brunot V, Besnard N, Benomar R, Daubin D, Ceballos P, Rispail P, Lachaud L, Bourgeois N, Klouche K. Emerging Invasive Fungal Infections in Critically Ill Patients: Incidence, Outcomes and Prognosis Factors, a Case-Control Study. J Fungi (Basel). 2021 Apr 24;7(5):330. doi: 10.3390/jof7050330. PMID 33923333